CLINICAL TRIAL: NCT07316881
Title: Acute Effects of an Elastic Band Warm-Up Protocol on Sprint and Vertical Jump Performance in Highly Trained Female Football Players
Brief Title: Effects of an Elastic Band Warm-Up on Sprint and Vertical Jump Performance in Female Football Players
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Institute of Maia (Other)
Responsible Party: Principal Investigator, Henrique Sousa, Principal Investigator, University Institute of Maia
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: EBT_HS_03
Record Dates: First submitted 2025-12-09; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Physical Performance Parameters

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standardized Warm-Up (WU) (Experimental): The standard active WU will consist of a brief aerobic portion, dynamic stretching, post-activation exercises and sprints/race-pace efforts.
  Interventions: Other: Standardized Warm-Up
- Warm-Up + Elastic Band (WU + EB) (Experimental): Participants will complete the standardized warm-up routine followed immediately by an elastic band activation protocol using looped resistance bands.
  Interventions: Other: Standardized Warm-Up; Other: Elastic Band Exercises
- Elastic Band + Warm-Up (EB + WU) (Experimental): Participants first perform the elastic band protocol using looped resistance bands. Immediately afterward, they complete the standardized warm-up routine.
  Interventions: Other: Standardized Warm-Up; Other: Elastic Band Exercises

INTERVENTIONS:
Other: Standardized Warm-Up — 2 minutes jogging and 4x30m side run; dynamic stretching for main locomotive lower limb muscles (2x10 hip adduction, 2x10 hip abduction, 2x10 butt kicks, 2x10 knee raises and 2x10 straight leg march), dynamic strength exercises (2x10 deep squats, and 2x10 forward lunges); incremental intermittent sprints and agility runs as follow: 2x10m pace, 2x20m pace, 2x30m pace, 1x30m with 10 decelerations (both feet), 1x30m with 10 decelerations (one foot), 2x30m with 4 changes of direction pace (90˚), 1x20m full pace and 1x30m full pace. The total time ofthe WU will be approximately 15 minutes.
Other: Elastic Band Exercises — Squats (10 reps), Hip Flexion (10 reps, each leg), Hip Extension (10 reps, each leg), Hip Abduction (10 reps, each leg), Hip Flexion with Knee Flexion (10 reps, each leg), Cross Walks (10 reps, forth and back) (All exercises are with elastic bands looped around the lower limbs)
  Arms: Elastic Band + Warm-Up (EB + WU); Warm-Up + Elastic Band (WU + EB)

SUMMARY:
This study aims to examine the acute effects of an elastic band warm-up on sprinting and vertical jump performance in female football players. A crossover design will be used across three separate sessions: (1) standardized warm-up (WU), (2) warm-up followed by elastic band activation (WU + EB), and (3) elastic band activation followed by the warm-up (EB + WU).

Performance evaluations-including sprint time and vertical jump height and power-will be conducted at three time points during each session: baseline (before the warm-up), immediately after the warm-up intervention, and 10 minutes post-intervention. This structure will allow the study to compare the immediate and short-term effects of different warm-up sequences involving elastic bands on neuromuscular performance. The findings may help optimize warm-up strategies to enhance acute athletic performance in female football players.

ELIGIBILITY:
Inclusion Criteria:

* belong to the U-19 or Senior level of a women's football (soccer) club.
* be apart of a national football championship

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Biologically Female
Enrollment: 22 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Vertical jump | The evaluations will be conducted at baseline (before the warm-up), immediately after the warm-up intervention, and 10 minutes post-intervention.
  Jump height and power will be evaluated using force plates (ForceDecks, Vald). The players will perform the countermovement jump, where they will begin from an upright position; a rapid downward movement to a knee angle of ∼90°, immediately transitioning to propel themselves upwards into the air.
Sprint Speed | The evaluations will be conducted at baseline (before the warm-up), immediately after the warm-up intervention, and 10 minutes post-intervention.
  Sprint performance will be measured over 10 m and 20 m using photocell timing gates (Microgate). Players will begin from a standardized starting position, with the front foot placed 50 cm behind the first timing gate. Upon their own cue, athletes will accelerate maximally through the course, ensuring consistent running mechanics while crossing both the 10-m and 20-m gates at full speed for accurate measurement of short-distance sprint times.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade da Maia, Porto, Maia, Portugal

IPD SHARING:
Plan to Share IPD: Undecided